CLINICAL TRIAL: NCT03782506
Title: The Impact of Music Therapy on Opioid Use in Cancer Survivors With Chronic Pain
Brief Title: Pain Management Support Study for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Joke Bradt, Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3R01NR016681-02S1 (NIH)
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Pain, Chronic; Opioid Use
Keywords: music therapy; pain management; opioid use; cancer survivors
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Music Therapy (Experimental): Ten 45-minute individual interactive music therapy sessions.
  Interventions: Behavioral: Interactive Music Therapy
- Verbal-based Support (Active Comparator): Ten 45-minute individual verbal support sessions.
  Interventions: Behavioral: Verbal-based support

INTERVENTIONS:
Behavioral: Interactive Music Therapy — Ten 45-minutes individual interactive music therapy (IMT) sessions delivered by a board-certified music therapist. Sessions start with music-guided breathing or humming. The music therapist then engages the participant in singing of familiar songs and co-created vocal or instrumental music improvisations. Discussion about the meaning assigned to songs and emotions expressed through the improvisations follow. Each session involves learning and practicing music-based techniques for the self-management of pain, anxiety, stress, mood, fatigue, and sleep disturbance as these are common opioid withdrawal symptoms. Psychoeducation about opioid tapering is provided and tapering challenges experienced by the patient will be actively addressed through music-based interventions.
  Arms: Interactive Music Therapy
Behavioral: Verbal-based support — Ten 45-minute individual sessions delivered by a master's level clinician with training in counseling. The sessions are focused on patient-initiated conversations about their pain, life stressors and the impact on their daily life. The intervener provides nondirective, supportive care by offering supportive, validating statements and reflective listening. The intervener refrains from employing active suggestion, problem-solving or behavioral or cognitive therapy techniques. The verbal support sessions are aimed at providing an empathic, therapeutic environment to facilitate emotional expression and sharing of worries and fears. As in the IMT protocol, psychoeducation about opioid tapering will be included and will be considered the only active treatment factor for this intervention.
  Arms: Verbal-based Support

SUMMARY:
Pain in cancer survivors is difficult to treat, and unrelieved pain can greatly reduce a person's quality of life. Opioids are often prescribed for pain management, yet they can have undesirable side effects and may put someone at risk for addiction or dependence. The purpose of this study is to examine the impact of an interactive music therapy intervention on pain management and opioid use in cancer survivors.

DETAILED DESCRIPTION:
As many as 40% of cancer survivors report experiencing chronic pain, and recent research indicates that pain is not well managed. Opioids are often prescribed during active cancer treatment for pain management, and many cancer survivors continue the same pain management regimen long after completing their cancer treatment. Reports indicate that prescription rates are up to 1.22 times higher for cancer cancer survivors than people without a cancer diagnosis, and the American Society of Clinical Oncology recommends that opioid tapering should be a priority once someone moves into survivorship status. Music interventions have been used for pain management in people with cancer, yet few studies have examined music therapy for chronic pain in cancer survivors. Moreover, none of these studies have not examined opioid use as a measure. Therefore, the overarching goals of this pilot study are to investigate the impact of an interactive music therapy (IMT) intervention on pain management and opioid use in cancer survivors with chronic pain versus a verbal-based support program (social attention control). This pilot study uses a mixed methods intervention design in which qualitative data (i.e. semi-structured follow-up interviews) are embedded within a randomized controlled trial. We will randomize 40 cancer survivors to one of two 10-session treatments: 1) Interactive Music Therapy or 2) Social Attention Control. Primary (mean daily opioid use) and secondary outcomes (pain intensity, pain interference, pain-related self-efficacy, patient perception of change, and physician perception of change in pain management) will be measured at baseline, post-intervention and 3-month follow-up. Follow-up interviews with a subsample of 12 participants and 4 physicians will enable us to gain a better understanding of potential treatment benefits, learn about challenges encountered, and obtain suggestions for treatment optimization. This is the first music therapy study to examine the benefits of music therapy for opioid tapering in cancer survivors with chronic pain and the results will be used to establish estimates of variance for sample size calculations for a larger-scale randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* adult cancer survivors
* chronic pain for ≥ 3 months
* chronic opioid use (i.e., use of opioids for more than 90 days)
* willingness to reduce the amount of opioids currently taking

Exclusion Criteria:

* history of polysubstance abuse/substance use disorder
* currently receiving methadone maintenance or suboxone treatment
* active psychosis or dementia
* inability to speak or write English
* moderate to severe hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Daily opioid dose | Through study completion, a maximum of 28 weeks
  Taking information from the Prescription Drug Monitoring Program, we will calculate the mean daily opioid dose for each participant by dividing the quantity of opioid pills prescribed by the number of days for which it was supplied.
Self-reported opioid use | Through study completion, a maximum of 28 weeks
  Self-report on intake of opioids and NSAIDS through daily pain medication log

SECONDARY OUTCOMES:
Pain intensity | At baseline, post-intervention (week 10), and 3-month follow up
  Measured by PROMIS® Pain Intensity-Short Form (SF)3a
Pain interference | At baseline, post-intervention (week 10), and 3-month follow up
  Measured by PROMIS® Cancer-Pain Interference -SF 6b
Self-efficacy | At baseline, post-intervention (week 10), and 3-month follow up
  Measured by PROMIS® Self-Efficacy of Symptoms
Patient perception of change | At post-intervention (week 10) and 3-month follow up
  Measured by Patient Global Impression of Change Scale (PGIC)
Physician perception of change | At baseline, post-intervention (week 10), and 3-month follow up
  A brief questionnaire asking about their perception of how the participant is doing in terms of pain management
Anxiety | At baseline, post-intervention (week 10), and 3-month follow up
  Measured by the PROMIS® Emotional Distress-Anxiety - SF6a
Depression | At baseline, post-intervention (week 10), and 3-month follow up
  Measured by the PROMIS® Depression - SF 6a
Sleep quality | At baseline, post-intervention (week 10), and 3-month follow up
  Measured by the PROMIS® Sleep Disturbance - SF4a

CONTACTS AND LOCATIONS:
Overall Officials: Joke Bradt, PhD, Principal Investigator — Drexel University
Locations (3):
- United States (3):
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Cancer Treatment Centers of America (CTCA), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
We will make the de-identified datasets available to other researchers. Researchers will be asked to submit a formal request for data sharing to the PI that outlines the purpose of the secondary data analysis. Data and associated documentation will be made available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol
Time Frame: After completion of study report and publication of the results
Access Criteria: We will make the de-identified datasets available to other researchers. Researchers will be asked to submit a formal request for data sharing to the PI that outlines the purpose of the secondary data analysis. Data and associated documentation will be made available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.